CLINICAL TRIAL: NCT05927168
Title: Effect of TENS Application After Thoracic Surgery on Pain Level and Analgesic Consumption During Breast Tube Extraction
Brief Title: Effect of TENS Application After Thoracic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Acelya Turkmen, PhD, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CU-SBF-AT-04
Record Dates: First submitted 2023-06-12; First posted 2023-07-03 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Transcutaneous Electrical Nerve Stimulation; Procedural Pain
MeSH Terms: conditions — Pain, Procedural | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TENS group (Experimental): TENS will be applied to the experimental group 45 minutes before the chest tube is removed and another 15 minutes after the chest tube is removed.
  Interventions: Device: TENS
- Control group (No Intervention): TENS will not be applied to the control group

INTERVENTIONS:
Device: TENS — TENS will be applied to the experimental group 45 minutes before the chest tube is removed and another 15 minutes after the chest tube is removed. Patients' pain scores will be evaluated using the Numerical Pain Scale (SAS) just before the TENS procedure, while the chest tube is removed, and 5 minutes after the TENS application is finished.
  Arms: TENS group

SUMMARY:
After thoracic surgery, a chest tube is inserted to evacuate the air and fluid formed in the pleural space and to provide hemodynamic stability. During chest tube placement, subcutaneous tissue layers, muscles and parietal pleura are passed through. This process is a trauma and the affected tissues show an inflammatory reaction to the trauma. The chest tube adheres to the tissue it comes into contact with and may experience mild, moderate and severe pain due to the separation of the adhesion due to pulling during removal. Chest tube removal is described as a severely painful procedure in studies. Analgesics are generally used in the treatment of acute pain during chest tube removal (Wei et al. 2022). However, pain guidelines and studies recommend the use of analgesics with non-pharmacological methods in order to minimize the pain experienced during chest tube removal and to provide adequate analgesia. One of the non-pharmacological methods used in pain management is Transcutaneous Electrical Nerve Stimulation (TENS). TENS, an electroanalgesia method, helps to control pain by providing skin stimulation through surface electrodes placed on the skin.While there are studies in the literature on the use of TENS in reducing the pain caused by chest tube removal after different surgical interventions, there are limited studies investigating the effect of TENS on the level of pain during chest tube removal and postoperative analgesic consumption after thoracic surgery. In this context, in this study, it is aimed to determine the effect of TENS application after thoracic surgery on pain level and analgesic requirement during chest tube removal.

DETAILED DESCRIPTION:
One of the non-pharmacological methods used in pain management is Transcutaneous Electrical Nerve Stimulation (TENS). Nurses play an important role in patient follow-up after surgery. It also has the responsibility to administer analgesics with the least side effects and the most effect. The New York Association of Nurses states that TENS is a complementary treatment method and its application strengthens the professional independence of nurses. However, as a result of our studies and observations, it is seen that there is no protocol for the use of TENS after thoracic surgery. TENS is applied together with physicians according to the nursing regulations in Turkey. Postoperative pain management requires team collaboration. Therefore, nurses should play a key role in pain management and use non-pharmacological methods.

ELIGIBILITY:
Inclusion Criteria:

* be over 18 years old
* no chest tube
* not have a pacemaker or arrhythmia
* no history of pain, alcohol use or substance abuse
* no prior pre-operative TENS/opioid use
* no postoperative epidural analgesics
* no history of psychiatric illness
* no history of metastatic disease
* being conscious, able to speak
* no barriers to the application of TENS
* no postoperative complications and being I, II and III in the ASA classification of the American Society of Anesthesiology.

Exclusion Criteria:

* having a history of epilepsy
* using analgesics at least 1 hour before chest tube removal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in the pain level | 1 hour
  Reducing the pain level of patients by applying TENS. Patients' pain scores before, during and after the procedure will be evaluated using the VAS.
Change in analgesic consumption | 2 hour
  Reducing analgesic consumption of patients by applying TENS. The analgesic consumption in the first 2 hour after the procedure will be learned by using the questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Açelya Türkmen, PhD, Principal Investigator — Cukurova University
Locations (1):
- Cukurova University, Adana, Sarıcam, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No